CLINICAL TRIAL: NCT02292082
Title: The Combination of Adductor Canal Block and Periarticular Injection. A Novel Technique for Patients Undergoing Total Knee Replacement (ACB PAI)
Acronym: ACB PAI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-018
Record Dates: First submitted 2014-11-10; First posted 2014-11-17 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis
Keywords: Nerve Block; Rehabilitation; Knee Replacement, Total
MeSH Terms: conditions — Osteoarthritis | interventions — Bupivacaine; Morphine; Methylprednisolone; Cefazolin; Saline Solution; Midazolam; Propofol; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peri-Articular Injections only (Active Comparator): Intra-Operatively
  * Spinal anesthetic with 0.5% bupivacaine (10 or 12.5)
  * Surgeon will perform the periarticular injections:
  * First deep injection prior to cementation Bupivacaine 0.5% with epinephrine, 30cc Morphine, 8 mg/ml, 1 cc Methylprednisolone, 40 mg/ml, 1 ml Cefazolin, 500 mg in 10 ml Normal saline, 22cc
  * Second superficial injection prior to closure. 1.20 ml 0.25% bupivacaine
  * Intravenous sedation with midazolam and propofol.
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Methylprednisolone; Drug: Cefazolin; Drug: Normal saline; Drug: Midazolam; Drug: Propofol; Drug: Dexamethasone
- Peri-Articular Injections and Adductor Canal Block (Experimental): Intra-Operatively
  * Spinal anesthetic with 0.5% bupivacaine (10 or 12.5)
  * Adductor canal block technique:
  * Supine position, after IV sedation
  * Ultrasound guided with linear transducer 8 MHz. Chiba needle, 22 G / 4 inches
  * Femoral artery will be identified in the adductor canal deep to the Sartorius muscle
  * 15 cc of Bupivacaine 0.25% with 2 mg of Preservative free Dexamethasone
  * Local anesthetic will be delivered periarterial between 12 and 6 o'clock
  * Intravenous sedation with midazolam and propofol.
  * First deep injection prior to cementation Bupivacaine 0.5% with epinephrine, 30cc Morphine, 8 mg/ml, 1 cc Methylprednisolone, 40 mg/ml, 1 ml Cefazolin, 500 mg in 10 ml Normal saline, 22cc
  * Second superficial injection prior to closure. 20 ml 0.25% bupivacaine
  Interventions: Drug: Bupivacaine; Drug: Morphine; Drug: Methylprednisolone; Drug: Cefazolin; Drug: Normal saline; Drug: Midazolam; Drug: Propofol; Drug: Dexamethasone; Device: 8 MHz. Chiba needle, 22 G / 4 inches

INTERVENTIONS:
Drug: Bupivacaine
Drug: Morphine
Drug: Methylprednisolone
Drug: Cefazolin
Drug: Normal saline
Drug: Midazolam
Drug: Propofol
Drug: Dexamethasone
Device: 8 MHz. Chiba needle, 22 G / 4 inches
  Arms: Peri-Articular Injections and Adductor Canal Block

SUMMARY:
Total knee replacement is associated with severe post-operative pain. The purpose of this study is to compare two methods of treatment for pain control following Total Knee Replacement with an accelerated physical therapy protocol to aid the achievement of rehab milestones.

DETAILED DESCRIPTION:
A total of 106 patients undergoing total knee arthroplasty will be randomized into two groups: one to receive only Periarticular injections and the other periarticular injections AND adductor canal block.

Patients will be asked their numeric pain scores before surgery as baseline and at 24 and 48 hours post-operation. Patients also will be asked questions from painOUT questionnaire at 24 and 48 hours.

Time to reach discharge criteria based on physical therapy assessments will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled for primary tricompartmental total knee arthroplasty with a participating surgeon
* Age 18 to 80 years
* Planned use of regional anesthesia
* Ability to follow study protocol
* English speaking (secondary outcomes include questionnaires validated in English only)

Exclusion Criteria:

Hepatic or renal insufficiency Patients younger than 18 years old and older than 80 Patients intending to receive general anesthesia Patients planning to go to rehab post operatively Patients scheduled to go into the OR after 1 pm Allergy or intolerance to one of the study medications Patients with an ASA of IV Chronic gabapentin/pregabalin use (regular use for longer than 3 months) Chronic opioid use (taking opioids for longer than 3 months) Diabetes Patients on workers compensation or disability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique A Goytizolo, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Peri-Articular Injections Only: Intra-Operatively
  * Spinal anesthetic with 0.5% bupivacaine (10 or 12.5)
  * Surgeon will perform the periarticular injections:
  * First deep injection prior to cementation Bupivacaine 0.5% with epinephrine, 30cc Morphine, 8 mg/ml, 1 cc Methylprednisolone, 40 mg/ml, 1 ml Cefazolin, 500 mg in 10 ml Normal saline, 22cc
  * Second superficial injection prior to closure. 1.20 ml 0.25% bupivacaine
  * Intravenous sedation with midazolam and propofol.
  Bupivacaine
  Morphine
  Methylprednisolone
  Cefazolin
  Normal saline
  Midazolam
  Propofol
  Dexamethasone
- Peri-Articular Injections and Adductor Canal Block: Intra-Operatively
  * Spinal anesthetic with 0.5% bupivacaine (10 or 12.5)
  * Adductor canal block technique:
  * Supine position, after IV sedation
  * Ultrasound guided with linear transducer 8 MHz. Chiba needle, 22 G / 4 inches
  * Femoral artery will be identified in the adductor canal deep to the Sartorius muscle
  * 15 cc of Bupivacaine 0.25% with 2 mg of Preservative free Dexamethasone
  * Local anesthetic will be delivered periarterial between 12 and 6 o'clock
  * Intravenous sedation with midazolam and propofol.
  * First deep injection prior to cementation Bupivacaine 0.5% with epinephrine, 30cc Morphine, 8 mg/ml, 1 cc Methylprednisolone, 40 mg/ml, 1 ml Cefazolin, 500 mg in 10 ml Normal saline, 22cc
  * Second superficial injection prior to closure. 20 ml 0.25% bupivacaine
  Bupivacaine
  Morphine
  Methylprednisolone
  Cefazolin
  Normal saline
  Midazolam
  Propofol
  Dexamethasone
  8 MHz. Chiba needle, 22 G / 4 inches
Period: Overall Study
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Started | 56 | 55
Completed | 56 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.6) | 66.9 (6.6) | 65.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 23 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 54 | 51 | 105
  Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 44 | 46 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 56 | 55 | 111

OUTCOME MEASURES:

1. Primary Outcome: Time to Meet Physical Therapy Discharge Criteria
Description: Time to reach physical therapy (PT) goals
Time Frame: First 3 days post-operatively
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 56 | 55
Minutes | 2109.3 (1232.8) | 1883.1 (846.2)

2. Secondary Outcome: Numerical Rating Scale (NRS) Pain Scores With Ambulation Postoperative Day 1
Description: Patient reported pain scores on postoperative day 1 from 0-10. 0 being no pain, 10 being the worst pain imaginable.
Time Frame: 24 hours after operating room discharge
Population: Unable to gather outcome data from all patients due to various reasons (exclusions, withdrawals, logistical reasons)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 53 | 53
score on a scale | 4.3 (2.6) | 3.9 (2.6)

3. Secondary Outcome: NRS Pain Score With Movement POD2
Description: NRS pain with movement as reported by the patient. Rated from 0-10. 0 being no pain, 10 being the worst pain imaginable.
Time Frame: 48 hours after surgery
Population: Unable to gather outcome data from all patients due to various reasons (exclusions, withdrawals, discharge, logistical reasons)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 34 | 32
score on a scale | 4.7 (1.6) | 5.2 (2.1)

4. Secondary Outcome: Opioid Consumption Postoperative Day (POD) 1
Description: Opioid consumption for patients from 0-24 hours postoperative, measured in mg OME (oral morphine equivalents)
Time Frame: 0-24 hours postoperatively
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg OME
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 56 | 54
mg OME | 58.4 (37.8) | 47.5 (40.3)

5. Secondary Outcome: Opioid Consumption POD2
Description: Opioid consumption over hours 24-48 postoperatively. Measured in mg OME (oral morphine equivalents). Higher equates to more opioids consumed.
Time Frame: 24-48 hours postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg OME
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 41 | 37
mg OME | 67.9 (49.1) | 60.1 (48.8)

6. Secondary Outcome: Hospital Length of Stay
Description: Measured in minutes.
Time Frame: Average of 3 days
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 56 | 55
Minutes | 3491 (1151.7) | 3394.4 (945.2)

7. Secondary Outcome: Patient Outcome Questionnaire (painOUT) Least Pain for 0-24 Hours Postoperatively
Description: Measures: least pain in the last 24 hours. Scores are measured from 0-10. 0 being no pain to 10 being the worst pain imaginable.
Time Frame: Participants will be followed for the duration of 2 days post operatively in the hospital
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 55 | 55
score on a scale | 1.5 (1.8) | 0.8 (1.6)

8. Secondary Outcome: Patient Outcome Questionnaire (painOUT) Least Pain for 24-48 Hours Postoperatively
Description: Least pain experienced from 24-48 hours postoperative on a scale from 0-10. 0 being no pain at all to 10 being the worst pain imaginable
Time Frame: 24-48 hours postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 34 | 33
score on a scale | 1.7 (1.5) | 1.8 (1.5)

9. Secondary Outcome: Patient Outcome Questionnaire (painOUT) Most Pain for 0-24 Hours Postoperatively
Description: Painout most pain experienced 0-24 hours postoperatively, measured from 0-10. 0 being no pain to 10 being the worst pain imaginable
Time Frame: 0-24 hours postoperatively
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 53 | 52
score on a scale | 6.7 (2.5) | 5.3 (2.9)

10. Secondary Outcome: Patient Outcome Questionnaire (painOUT) Most Pain for 24-48 Hours Postoperatively
Description: Painout most pain experienced 24-48 hours postoperatively measured on a scale from 0-10. Higher scores indicate higher pain levels.
Time Frame: 24-48 hours postoperative
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 53 | 52
score on a scale | 6.9 (2.3) | 6.6 (2.3)

11. Secondary Outcome: Knee Society Score (KSS) at 6 Weeks Postoperatively
Description: KSS (Knee Society Score) score measured at 6 weeks postoperatively. The scale is from 0-100. Scores below 60 indicate poor function, 60-69 indicate fair, 70-79 indicate good, and 80-100 indicate excellent functional scores. KSS measures knee pain, flexion contracture,extension lag, alignment, stability, and total range of flexion and generates an associated score correlating to knee function. Higher is better. There is no sub score - only the cumulative Knee Society Score.
Time Frame: Post operatively at approximately 6 weeks after surgery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
Number analyzed (Participants) | 17 | 17
score on a scale | 85.2 (20) | 75.2 (17.7)

ADVERSE EVENTS:
Arm/Group | Peri-Articular Injections Only | Peri-Articular Injections and Adductor Canal Block
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55
Other Adverse Events (participants affected / at risk) | 0/56 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-03-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT02292082/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT02292082/Prot_SAP_001.pdf